CLINICAL TRIAL: NCT04236817
Title: Impact on Patient COmpliance With Medication Using Pre-packaged Blisters for Long-term Medical therapY
Acronym: I-COMPLY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: The Huron Foundation (Unknown)
Responsible Party: Principal Investigator, Andrei Brateanu, MD, MD, Principal Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 14-1554
Record Dates: First submitted 2019-12-19; First posted 2020-01-22 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Medication Adherence; Medication Compliance
Keywords: Medication Adherence; Medication compliance; Pill-packaging
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Intervention Model Description: Open label randomized controlled trial. The patient population included 114 patients, followed by primary care physicians at the Cleveland Clinic Stephanie Tubbs Jones Health Center, taking four or more medication doses daily. They were randomized either to the intervention group or the control group. Patients in the intervention group received prescriptions pre-packaged in individual packets that were delivered by the pharmacy. Patients in the control group continued to receive medications from pharmacies as they did prior to enrollment. The primary outcome was the percentage of missed pills in the intervention group versus the control group after four months of enrollment. The secondary outcome was the number of daily doses missed. The number and percentages of missed pills for each subject was calculated and summarized by group. The primary analysis compared the mean percentage of missed pills between the two groups using t-test analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-packed blisters for distribution of medications (Experimental): Patients in the intervention group received prescriptions pre-packaged in individual packets that were delivered by the pharmacy.
  Interventions: Behavioral: Pre-packed blisters for distribution of medications
- Routine distribution of medications (Placebo Comparator): Patients in the control group continued to receive medications from pharmacies as they did prior to enrollment.
  Interventions: Behavioral: Routine distribution of medications

INTERVENTIONS:
Behavioral: Pre-packed blisters for distribution of medications
  Arms: Pre-packed blisters for distribution of medications
Behavioral: Routine distribution of medications
  Arms: Routine distribution of medications

SUMMARY:
The use of packaging interventions like pillboxes or blister packs has been shown to significantly improve medication adherence. The purpose of this study is to assess the effect of home-delivered pill packs on medication adherence in a low-income population. This is an open-lab randomized controlled trial taking four or more medication doses daily, randomized either to the intervention group or the control group. Patients in the intervention group received prescriptions pre-packaged in individual packets that were delivered by the pharmacy. Patients in the control group continued to receive medications from pharmacies as they did prior to enrollment. The primary outcome was the percentage of missed pills in the intervention group versus the control group after four months of enrollment.

DETAILED DESCRIPTION:
For patients in the study group, new prescriptions with three refills were electronically scripted to local compliance packaging pharmacy, ExactCare pharmacy, LLC, Valley View, Ohio, 44125. ExactCare is a local packaging pharmacy that pre-packs medications for patients so that each day's medications come in a separate paper compartment that can be discarded after daily use. They also deliver medications to the patients' homes. At the initiation of the study, ExactCare provided medications in pill packs for all patient medications in a 30-day supply (Figure 2). Pill bottle medications were provided for medications that would run out prior to the initial supply date. Inhalers, nebulizers, injectable medications, as needed medications and medications that required frequent dose changes were not included in the pill packs but were sent separately within the 30-day supply box.

If the patient was started on a new medication by their PCP, the local compliance packaging pharmacy packed this medication in pill packs for the next 30-day box supply and sent pill bottles containing enough pills to last the patient till the next 30-day box. Every pill in the pill pack was coded with an identification number. If the patient's physician discontinued or changed the dose of any medication, the patient was advised to remove the pill from the pack using its identification number and either discard it or make the dose change accordingly.

A study investigator counted the pills left in the control group prior to the study start date. After the study start date, patients in the control group continued to receive their medications the same way they were getting them before being enrolled in this study using either electronic or printed prescriptions. They received instructions about the timing and frequency of medication administration from their physicians and nurses, and picked up their medications from their local pharmacy.

Patients from both groups had a follow-up PCP visit approximately four months from enrollment. Patients received telephone calls prior to their follow-up appointments to remind them to bring their medications from home. During the appointment, the study investigator counted the medications remaining in the pill packs for the study group patients and the pills remaining in pill bottles for the control group patients.

ExactCare provided the initial start date for each patient receiving their pill packs in 30-day supply. Refill dates were accessed from local pharmacies and the EMR for patients in the control group. This information was used to calculate the number of pills expected to remain with each patient at the end of the study and to compare to the actual number of pills remaining. New medications, discontinued medications, and modified-dose medications were not included in the study analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or older
* Covered by Medicaid insurance
* Seen in clinic at least two times within the past year, follow-up appointment scheduled between January and May 2015
* Prescribed a minimum of four medications daily

Exclusion Criteria:

* Nursing home patients
* Patients with planned hospital stays during the study period
* Patients who were already receiving medications in pre-packed blisters or pill packs prior to study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2015-05-30 (Actual); Study Completion 2015-05-30 (Actual)

PRIMARY OUTCOMES:
Percentage of missed pills | 4 month follow-up
  The primary outcome was the percentage of missed pills in the intervention group versus the control group after four months of enrollment.

SECONDARY OUTCOMES:
Percentage of missed doses | 4 month follow-up
  The secondary outcome was the number of daily doses missed.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ward BW, Schiller JS, Goodman RA. Multiple chronic conditions among US adults: a 2012 update. Prev Chronic Dis. 2014 Apr 17;11:E62. doi: 10.5888/pcd11.130389. PMID 24742395
- [Background] Ward BW, Schiller JS. Prevalence of multiple chronic conditions among US adults: estimates from the National Health Interview Survey, 2010. Prev Chronic Dis. 2013 Apr 25;10:E65. doi: 10.5888/pcd10.120203. PMID 23618545
- [Background] Blazing MA, Giugliano RP, Cannon CP, Musliner TA, Tershakovec AM, White JA, Reist C, McCagg A, Braunwald E, Califf RM. Evaluating cardiovascular event reduction with ezetimibe as an adjunct to simvastatin in 18,144 patients after acute coronary syndromes: final baseline characteristics of the IMPROVE-IT study population. Am Heart J. 2014 Aug;168(2):205-12.e1. doi: 10.1016/j.ahj.2014.05.004. Epub 2014 May 15. PMID 25066560
- [Background] A Randomized Trial of Intensive versus Standard Blood-Pressure Control. N Engl J Med. 2017 Dec 21;377(25):2506. doi: 10.1056/NEJMx170008. No abstract available. PMID 29262284
- [Background] Sabatine MS, Giugliano RP, Wiviott SD, Raal FJ, Blom DJ, Robinson J, Ballantyne CM, Somaratne R, Legg J, Wasserman SM, Scott R, Koren MJ, Stein EA; Open-Label Study of Long-Term Evaluation against LDL Cholesterol (OSLER) Investigators. Efficacy and safety of evolocumab in reducing lipids and cardiovascular events. N Engl J Med. 2015 Apr 16;372(16):1500-9. doi: 10.1056/NEJMoa1500858. Epub 2015 Mar 15. PMID 25773607
- [Background] Pasina L, Brucato AL, Falcone C, Cucchi E, Bresciani A, Sottocorno M, Taddei GC, Casati M, Franchi C, Djade CD, Nobili A. Medication non-adherence among elderly patients newly discharged and receiving polypharmacy. Drugs Aging. 2014 Apr;31(4):283-9. doi: 10.1007/s40266-014-0163-7. PMID 24604085
- [Background] Marcum ZA, Gellad WF. Medication adherence to multidrug regimens. Clin Geriatr Med. 2012 May;28(2):287-300. doi: 10.1016/j.cger.2012.01.008. PMID 22500544
- [Background] Conn VS, Ruppar TM, Chan KC, Dunbar-Jacob J, Pepper GA, De Geest S. Packaging interventions to increase medication adherence: systematic review and meta-analysis. Curr Med Res Opin. 2015 Jan;31(1):145-60. doi: 10.1185/03007995.2014.978939. Epub 2014 Nov 4. PMID 25333709
- [Background] Osterberg L, Blaschke T. Adherence to medication. N Engl J Med. 2005 Aug 4;353(5):487-97. doi: 10.1056/NEJMra050100. No abstract available. PMID 16079372
- [Background] Ritchey M, Chang A, Powers C, Loustalot F, Schieb L, Ketcham M, Durthaler J, Hong Y. Vital Signs: Disparities in Antihypertensive Medication Nonadherence Among Medicare Part D Beneficiaries - United States, 2014. MMWR Morb Mortal Wkly Rep. 2016 Sep 16;65(36):967-76. doi: 10.15585/mmwr.mm6536e1. PMID 27632693
- [Background] Viswanathan M, Golin CE, Jones CD, Ashok M, Blalock SJ, Wines RC, Coker-Schwimmer EJ, Rosen DL, Sista P, Lohr KN. Interventions to improve adherence to self-administered medications for chronic diseases in the United States: a systematic review. Ann Intern Med. 2012 Dec 4;157(11):785-95. doi: 10.7326/0003-4819-157-11-201212040-00538. PMID 22964778
- [Background] Stuart B, Davidoff A, Lopert R, Shaffer T, Samantha Shoemaker J, Lloyd J. Does medication adherence lower Medicare spending among beneficiaries with diabetes? Health Serv Res. 2011 Aug;46(4):1180-99. doi: 10.1111/j.1475-6773.2011.01250.x. Epub 2011 Mar 17. PMID 21413981
- [Background] Stuart BC, Dai M, Xu J, Loh FH, S Dougherty J. Does good medication adherence really save payers money? Med Care. 2015 Jun;53(6):517-23. doi: 10.1097/MLR.0000000000000360. PMID 25961659
- [Background] Wroe AL. Intentional and unintentional nonadherence: a study of decision making. J Behav Med. 2002 Aug;25(4):355-72. doi: 10.1023/a:1015866415552. PMID 12136497
- [Background] Gerber BS, Cho YI, Arozullah AM, Lee SY. Racial differences in medication adherence: A cross-sectional study of Medicare enrollees. Am J Geriatr Pharmacother. 2010 Apr;8(2):136-45. doi: 10.1016/j.amjopharm.2010.03.002. PMID 20439063
- [Background] Lafata JE, Karter AJ, O'Connor PJ, Morris H, Schmittdiel JA, Ratliff S, Newton KM, Raebel MA, Pathak RD, Thomas A, Butler MG, Reynolds K, Waitzfelder B, Steiner JF. Medication Adherence Does Not Explain Black-White Differences in Cardiometabolic Risk Factor Control among Insured Patients with Diabetes. J Gen Intern Med. 2016 Feb;31(2):188-195. doi: 10.1007/s11606-015-3486-0. PMID 26282954
- [Background] Bahrami H, Kronmal R, Bluemke DA, Olson J, Shea S, Liu K, Burke GL, Lima JA. Differences in the incidence of congestive heart failure by ethnicity: the multi-ethnic study of atherosclerosis. Arch Intern Med. 2008 Oct 27;168(19):2138-45. doi: 10.1001/archinte.168.19.2138. PMID 18955644
- [Background] Lloyd-Jones D, Adams RJ, Brown TM, Carnethon M, Dai S, De Simone G, Ferguson TB, Ford E, Furie K, Gillespie C, Go A, Greenlund K, Haase N, Hailpern S, Ho PM, Howard V, Kissela B, Kittner S, Lackland D, Lisabeth L, Marelli A, McDermott MM, Meigs J, Mozaffarian D, Mussolino M, Nichol G, Roger VL, Rosamond W, Sacco R, Sorlie P, Stafford R, Thom T, Wasserthiel-Smoller S, Wong ND, Wylie-Rosett J; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Executive summary: heart disease and stroke statistics--2010 update: a report from the American Heart Association. Circulation. 2010 Feb 23;121(7):948-54. doi: 10.1161/CIRCULATIONAHA.109.192666. No abstract available. PMID 20177011
- [Background] Pi-Sunyer FX. Obesity and diabetes in blacks. Diabetes Care. 1990 Nov;13(11):1144-9. doi: 10.2337/diacare.13.11.1144. PMID 2261835
- [Background] Braverman J, Dedier J. Predictors of medication adherence for African American patients diagnosed with hypertension. Ethn Dis. 2009 Autumn;19(4):396-400. PMID 20073139
- [Background] Siegel D, Lopez J, Meier J. Antihypertensive medication adherence in the Department of Veterans Affairs. Am J Med. 2007 Jan;120(1):26-32. doi: 10.1016/j.amjmed.2006.06.028. PMID 17208076
- [Background] Williams A, Manias E, Walker R. Interventions to improve medication adherence in people with multiple chronic conditions: a systematic review. J Adv Nurs. 2008 Jul;63(2):132-43. doi: 10.1111/j.1365-2648.2008.04656.x. PMID 18537843
- [Background] Haynes RB, McDonald H, Garg AX, Montague P. Interventions for helping patients to follow prescriptions for medications. Cochrane Database Syst Rev. 2002;(2):CD000011. doi: 10.1002/14651858.CD000011. PMID 12076376
- [Background] Conn VS, Ruppar TM. Medication adherence outcomes of 771 intervention trials: Systematic review and meta-analysis. Prev Med. 2017 Jun;99:269-276. doi: 10.1016/j.ypmed.2017.03.008. Epub 2017 Mar 16. PMID 28315760
- See also: Health US, 2013 With Special Feature on Prescription Drugs — https://www.cdc.gov/nchs/data/hus/hus13.pdf

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-11-24): https://cdn.clinicaltrials.gov/large-docs/17/NCT04236817/Prot_SAP_000.pdf